CLINICAL TRIAL: NCT06517641
Title: A Phase II Trial of Non-Myeloablative Conditioning and Transplantation of Haploidentical Related, Partially HLA-Mismatched, or Matched Unrelated Bone Marrow for Newly Diagnosed Patients With Severe Aplastic Anemia
Brief Title: Clinical Trial of Upfront Haploidentical or Unrelated Donor BMT to Restore Normal Hematopoiesis in Aplastic Anemia
Acronym: BMT CTN CureAA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 2207; BMT CTN Protocol 2207 (Other: BMT CTN)
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Intervention Model Description: This is a parallel cohort study comprised of two cohorts - patients receiving haploidentical donor transplant and patients receiving unrelated donor transplant. The goal is 60 participants in total who initiate the protocol-specified conditioning regimen, 30 in each of the haploidentical and unrelated donor transplant cohorts. Additional participants may be screened, consented, and registered in order to reach accrual goals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Haploidentical transplantation (Active Comparator): Patients receiving bone marrow transplanted from a haploidentical related donor will be included in this arm.
  Interventions: Drug: Haploidentical donor bone marrow transplant
- Unrelated donor transplantation (Active Comparator): Patients receiving bone marrow transplanted from an unrelated donor will be included in this arm.
  Interventions: Drug: Unrelated donor bone marrow transplant

INTERVENTIONS:
Drug: Haploidentical donor bone marrow transplant — Drugs:
  1. Antithymocyte Globulin (ATG) dose will be 0.5 mg/kg IV on Day -9 over 6 hours and 2 mg/kg IV on Days -8 and -7 over 4 hours.
  2. Fludarabine dose will be 30 mg/m^2 IV daily for 5 days from Day -6 to Day -2.
  3. Cyclophosphamide dose will be 14.5 mg/kg IV daily for 2 days (Day -6 to Day -5) prior to transplantation and 50 mg/kg IV daily for 2 days (Day +3 to Day +4) after transplantation.
  4. Tacrolimus should be started on Day +5 and administered to maintain a level of 10-15 ng/mL.
  5. Mycophenolate mofetil (MMF) dose will be 15 mg/kg PO three times a day (TID) up to 1 gm TID (or IV equivalent) starting on Day +5 through Day +35.
  6. G-CSF will be given IV or SQ starting on Day +5 at 5 mcg/kg/day until ANC is > 1500 for 3 days.
  Radiation:
  1. Total Body Irradiation (TBI): will be given as a single dose of 400 cGy on Day -1.
  Procedure:
  1. HSCT: Eligible patients will receive a haploidentical donor bone marrow transplant.
  Arms: Haploidentical transplantation
Drug: Unrelated donor bone marrow transplant — Drugs:
  1. Antithymocyte Globulin (ATG) dose will be 0.5 mg/kg IV on Day -9 over 6 hours and 2 mg/kg IV on Days -8 and -7 over 4 hours.
  2. Fludarabine dose will be 30 mg/m^2 IV daily for 5 days from Day -6 to Day -2.
  3. Cyclophosphamide dose will be 14.5 mg/kg IV daily for 2 days (Day -6 to Day -5) prior to transplantation and 50 mg/kg IV daily for 2 days (Day +3 to Day +4) after transplantation.
  4. Tacrolimus should be started on Day +5 and administered to maintain a level of 10-15 ng/mL.
  5. Mycophenolate mofetil (MMF) dose will be 15 mg/kg PO three times a day (TID) up to 1 gm TID (or IV equivalent) starting on Day +5 through Day +35.
  6. G-CSF will be given IV or SQ starting on Day +5 at 5 mcg/kg/day until ANC is > 1500 for 3 days.
  Radiation:
  1. Total Body Irradiation (TBI): will be given as a single dose of 400 cGy on Day -1.
  Procedure:
  1. HSCT: Eligible patients will receive an unrelated donor bone marrow transplant.
  Arms: Unrelated donor transplantation

SUMMARY:
BMT CTN 2207 will investigate the use of marrow transplantation for treatment of severe aplastic anemia that has not previously been treated.

DETAILED DESCRIPTION:
This study is a prospective, multicenter Phase II study of hematopoietic stem cell transplantation for previously untreated patients with severe aplastic anemia (SAA). Severe Aplastic Anemia (SAA) is a rare condition in which the body stops producing enough new blood cells. Patients with aplastic anemia have low white blood cells (cells which fight infection), low red blood cells (cells that carry oxygen throughout the body), and low platelets (cells that help form clots and prevent bleeding). Treatments for SAA seeks to repair this abnormal immune system attack and allow the bone marrow to make the normal amount of blood cells. This can be done with a bone marrow transplant or with medications to suppress the immune system.

Historically, transplant therapy for SAA has been reserved for patients under 40 years old who had an available fully matched related donor. The standard treatment for older patients with SAA and patients who do not have a fully matched related donor has been treatment using transfusions, medications that suppress the immune system (immunosuppressive therapy, IST), and medications that try to stimulate the bone marrow to produce more cells. For these patients, transplant was used only if a patient did not respond to these interventions. However, progress has made transplantation safer and allowed for half-matched related donor or full or partially-matched unrelated donors to be used with success rates similar to fully matched related donors in many situations. The goals of this study are to determine if patients with SAA who have not received previous treatment for SAA can be treated effectively with transplant as their first SAA therapy.

This is a parallel cohort study comprised of two cohorts based on donor selection: haploidentical related donors and unrelated donors. The accrual goal is 30 participants enrolled and starting protocol-specified conditioning in each cohort, yielding 60 participants in total. Participants will be treated with a reduced-intensity preparative regimen of fludarabine (150 mg/m2), cyclophosphamide (29 mg/kg), low dose total body irradiation (TBI, 400 cGy), and Thymoglobulin® (4.5 mg/kg). Bone marrow will be collected from donors and fresh (not cryopreserved) cells will be given to patients. GVHD prophylaxis will be with post-HSCT cyclophosphamide (100 mg/kg), tacrolimus, and mycophenolate mofetil (MMF). All patients will receive the same conditioning regimen and GVHD prophylaxis. Participants will be followed for 1 year post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3 years to 75 years
2. Confirmed diagnosis of acquired SAA defined as:

   a. Bone marrow cellularity < 25% or variable marrow cellularity but with < 30% residual hematopoietic cells deemed HYPOcellular for age AND b. Two (2) out of 3 of the following (in peripheral blood). i. Neutrophils < 0.5 x109/L ii. Platelets < 20 x109/L iii. Reticulocyte count < 20 x109/L (< 60 x 109/L using an automated analysis)
3. No suitable fully matched related donor as per Investigator's discretion (6/6 match for HLA A and B at intermediate or high-resolution and DRB1 at high-resolution using deoxyribonucleic acid [DNA]-based typing) available.
4. Available donor as defined in the protocol.
5. Participant and/or legal guardian must sign informed consent.
6. Adequate organ function defined by institutional transplant standards or defined as below:

   1. Cardiac: Left ventricular ejection fraction (LVEF) at rest > 40% with no clinical signs of cardiac failure. For participants aged < 13 years, shortening fraction (SF) ≥ 26% by echocardiogram or multigated acquisition (MUGA) may be substituted for LVEF.
   2. Hepatic: Total bilirubin < 2.0 mg/dL unless Gilbert's disease is present
   3. Renal: For participants > 13.0 years of age at the time of enrollment: estimated creatinine clearance (CrCl) > 60 mL/minute (per institutional standard). For participants < 13.0 years of age at enrollment: glomerular filtration rate (GFR) estimated by the updated Schwartz formula ≥ 90 mL/min/1.73 m2. If the estimated GFR is < 90 mL/min/1.73 m2, then renal function must be measured by 24-hour creatinine clearance or nuclear GFR, and must be > 50 mL/min/1.73 m2.
   4. Pulmonary:

   i. For participants > 13.0 years of age: Diffusing capacity of the lung for carbon monoxide (DLCO, corrected/adjusted for hemoglobin [Hb]) > 50%, or Spirometry with forced expiratory volume 1 (FEV1) > 50% predicted (without administration of bronchodilator) and forced vital capacity (FVC) > 50% predicted.

   ii. For participants < 13.0 years of age unable to perform pulmonary function tests (PFTs) due to age or developmental ability: (1) no evidence of dyspnea at rest and (2) no need for supplemental oxygen and (3) O2 saturation > 92% on room air at sea level (with lower levels allowed at higher elevations per established center standard of care [e.g., Utah, 4,200 feet above sea level, does not give supplemental oxygen unless below 90%]).
7. Karnofsky or Lansky performance status ≥ 60%.
8. Females and males of childbearing potential must agree to practice 2 effective methods of contraception at the same time or agree to abstinence.

Exclusion Criteria:

1. Inherited bone marrow failure syndromes such as Fanconi anemia and short telomere syndromes must be ruled out according to center standards. It is recommended that functional testing for Fanconi Anemia (di-epoxybutane [DEB] chromosomal breakage analysis) and telomere length assessment be performed. If available, genetic panels for inherited bone marrow failure syndromes can be considered as an alternative to functional testing.
2. Clonal cytogenetic abnormalities consistent with pre-MDS or MDS on marrow examination (e.g., monosomy 7 and other MDS-defining changes per recent pathology guidelines).
3. Formal diagnosis of MDS by World Health Organization (WHO) 2022 or International Consensus Classification (ICC).
4. Recipient positive for HLA antibodies against a mismatched HLA in the selected donor determined by the presence of donor specific HLA antibodies (DSA) to any mismatched HLA allele/antigen at any of the following loci (HLA-A, -B, -C, -DRB1, DRB3, DRB4, DRB5, -DQA1, -DQB1, -DPA1, -DPB1) with median fluorescence intensity (MFI) >3000 by microarray-based single antigen bead testing. In patients receiving red blood cell or platelet transfusions, DSA evaluation must be performed or repeated post-transfusion and immediately prior to initiation of recipient preparative regimen to ensure there is confirmation of no DSA to the selected donor when conditioning starts.
5. Prior desensitization attempt for HLA antibodies to chosen donor. Any intervention with the sole intent to reduce the level of HLA DSA, (e.g., plasmapheresis, intravenous immunoglobulin [IVIG], MMF, etc.) would constitute a desensitization attempt.
6. Prior treatment for SAA (e.g., immunosuppressive therapy using ATG, calcineurin inhibitors [CNIs], thrombopoietin receptor agonists or androgens). Short courses of steroids or IVIG that were not explicitly administered for SAA therapy will be allowed.
7. Prior allogeneic stem cell transplant.
8. Prior solid organ transplant.
9. Known life-threatening reaction (i.e., anaphylaxis) to Thymoglobulin® (Sanofi) that would prohibit use for the participant as this study requires use of the Thymoglobulin® (Sanofi) preparation of ATG.
10. Uncontrolled bacterial, viral, or fungal infection at the time of enrollment. Uncontrolled is defined as currently taking medication and with progression or no clinical improvement on adequate medical treatment.
11. Female participants who are pregnant, as detected using a pregnancy test as per institutional practice, or breast-feeding.
12. Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent > 5 years previously will be allowed. Cancer treated with curative intent ≤ 5 years previously will not be allowed unless approved by the Protocol Chairs and/or Protocol Officer.

Of note, participants with seropositivity for the human immunodeficiency virus (HIV) may be considered if viral load is undetectable. Similarly, carriers of hepatitis B (HepB) or hepatitis C (HepC) may not have a detectable viral load of HepB virus or HepC virus.

Participants with HIV that is well-controlled on combination antiretroviral therapy and no AIDS related complications within the past 12 months are eligible.

Infections other than HIV:

* Prior infections must be controlled
* HepB participants are eligible if on effective suppressive therapy and otherwise meet inclusion/exclusion criteria
* HepC participants are eligible if otherwise meet inclusion/exclusion criteria

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Graft versus host disease (GVHD)-free failure-free survival (GFFS) at One year | 1 year after initiation of conditioning
  The primary endpoint is GFFS at 1 year after initiation of conditioning. Events for GFFS include Grade III-IV aGVHD, cGVHD requiring immunosuppression, primary or secondary graft failure requiring second definitive therapy, failure to receive an HSCT infusion, and death. GFFS is defined as the time interval from start of conditioning until the first of these events occurs. For failure to receive an HSCT infusion, the date will be at the time the decision not to proceed to HSCT is made.

SECONDARY OUTCOMES:
Percentage of Participants with Overall survival (OS) at One year post conditioning | 1 year after initiation of conditioning
  Events for OS include death from any cause. OS is defined as the time interval from initiation of conditioning until death. The OS probability will be assessed at 1 year after initiation of conditioning.
Percentage of Participants with Failure-Free Survival (FFS) at One year post conditioning | 1 year after initiation of conditioning
  Events for FFS include treatment failure or death. Treatment failure is defined as the initiation of treatment with a second definitive therapy. FFS is defined as the time interval from start of conditioning until the start date of a second definitive therapy or death, whichever occurs first.
Participants Alive and Engrafted at One year post conditioning | 1 year after initiation of conditioning
  The proportion of patients who are alive with donor cells present at 1 year after initiation of conditioning will be described, where the presence of donor cells is defined as achieving at least 5% myeloid donor chimerism (whole blood or marrow) in the most recent measurement through 1 year.
Percentage of Participants with Neutrophil Recovery post-transplant | Day 28 and Day 56 post-HSCT
  Neutrophil recovery is achieving an ANC ≥ 0.5 x109/L for 3 consecutive measurements on different days, with the first of the 3 days being defined as the day of neutrophil recovery. The cumulative incidences of neutrophil recovery at Day +28 and Day +56 post-HSCT will be estimated.
Percentage of Participants with Red Blood Cell Recovery post-transplant | Day 100, Day 180, and Day 365 post-HSCT
  Red blood cell (RBC) recovery is defined as Hb level ≥ 7 g/dL with no red cell transfusion in the preceding 7 days. The first day of the 7 days will be defined as the day of RBC recovery. The cumulative incidences of RBC recovery at Day +100, Day +180, and Day +365 post-HSCT will be estimated.
Percentage of Participants with Platelet Recovery post-transplant | Day 100 post-HSCT
  Platelet recovery is defined by achieving a platelet count ≥ 20 x 109/L with no platelet transfusions in the preceding 7 days. The first 7 days of the sustained platelet count will be defined as the day of platelet recovery. The cumulative incidence of platelet recovery at Day +100 post-HSCT will be estimated.
Percentage of Participants with Primary Graft Failure post-transplant | Day 56 post-HSCT
  * Primary Graft Failure is defined as the occurrence of any of the following:
    1. Lack of neutrophil recovery by Day +56 post-HSCT.
    2. Failure to achieve at least 5% myeloid donor chimerism any measurement up to and including Day +56 post-HSCT.
    3. Administration of a second definitive therapy, which is defined as a second transplant or a course of ATG.
  * The proportion of patients with primary graft failure through Day +56 post-HSCT will be estimated.
Percentage of Participants with Secondary Graft Failure post-transplant | 1 year post-HSCT
  * Secondary Graft Failure is defined as the occurrence of any of the following:
    1. Initial neutrophil recovery with donor chimerism greater than or equal to 5%, followed by sustained subsequent decline in ANC with donor chimerism declining to less than 5%.
    2. Administration of a second definitive therapy, which is defined as a second transplant or a course of ATG.
  * The cumulative incidence of secondary graft failure at 1 year post-HSCT will be estimated.
Percentage of Participants with any Graft Failure (primary or secondary) post-transplant | 1 year post-HSCT
  The time from transplant until any graft failure (primary or secondary) will be described for each transplant cohort using the Aalen-Johansen estimator, with death treated as a competing risk. Estimates and 90% CIs of the cumulative incidence of any graft failure will be provided at Day +365 post-HSCT for each cohort.
Participants with Hematologic Response post-transplant | Day 100, Day 180, and Day 365 post-HSCT
  Hematologic response will be assessed according to the modified NIH criteria determined at Day +100, Day +180, and Day +365 post-HSCT. Complete response (CR) is defined as meeting all 3 peripheral blood count criteria: 1) ANC > 1x 109/L; 2) Hb > 10g/dL; and 3) platelet count > 100 x 109/L. Partial response (PR) is defined as blood counts no longer satisfying criteria for SAA and having transfusion independence (defined as no need for packed red blood cell [PRBC] or platelet transfusions) but insufficient for a CR.
Percentage of participants with Grades II-IV and III-IV Acute GVHD at Day 100 post-transplant | Day 100 post-HSCT
  Acute GVHD was graded according to the BMT CTN Technical Manual of Operating Procedures (MOP) which describes the Mount Sinai Acute GVHD International Consortium (MAGIC). Higher GVHD grade indicates worse outcomes. Grade I is defined as Skin stage 1-2 and stage 0 for both GI and liver. Grade II is stage 3 skin, stage 1 GI, or stage 1 liver. Grade III is stage 2-3 GI or stage 2-3 liver. Grade IV is stage 4 skin or stage 4 liver. The cumulative incidences of Grade II-IV and Grade III-IV acute GVHD at Day +100 post-HSCT will be estimated.
Percentage of participants with Chronic GVHD at One year post-transplant | Day 365 post-HSCT
  Chronic GVHD are graded according to the BMT CTN Technical Guideline. The cumulative incidences of all chronic GVHD and of chronic GVHD requiring immunosuppression will be estimated.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Blood and Marrow Transplant Center at Northside Hospital, Atlanta, Georgia
  - University of Kansas Medical Center, Westwood, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, Barnes-Jewish Hospital, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to the NIH data and specimen central repository (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol
Time Frame: Within 6 months of official study closure at participating sites
Access Criteria: Available to public

REFERENCES:
- See also: Blood and Marrow Transplant Clinical Trials Network Website — http://bmtctn.net/

DOCUMENTS (5):
  • Study Protocol (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT06517641/Prot_000.pdf
  • Informed Consent Form: Assent to Participate in Research (12 to 17 years of age) (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT06517641/ICF_001.pdf
  • Informed Consent Form: Assent to Participate in Research (7 to 11 years of age) (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT06517641/ICF_002.pdf
  • Informed Consent Form: Haploidentical Donor Informed Consent (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT06517641/ICF_003.pdf
  • Informed Consent Form: Patient Informed Consent (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT06517641/ICF_004.pdf